CLINICAL TRIAL: NCT06713512
Title: invEstigating oeStrogen Signalling and the Effect upoN the exTracelluar Matrix In pAtients With Obstructive Lung Disease
Acronym: ESSENTIAL
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 326236
Record Dates: First submitted 2024-09-13; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Lung Disease; Respiratory Ilness; Estrogen Deficiency; Asthma
Keywords: Asthma; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with physician-diagnosed disease (Asthma and/or COPD).: People with physician-diagnosed disease (Asthma and/or COPD).
  Interventions: Other: No intervention
- Healthy controls: People with no physician-diagnosed disease (Asthma and/or COPD).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Intervention

SUMMARY:
This study aims to understand the role of oestrogen in patients with asthma and Chronic Obstructive Pulmonary Disorder (COPD). Therefore, what is the effect of oestrogen in these participants compared to controls (those without disease). The study hypothesises that oestrogen loss in patients with asthma and COPD causes accelerated lung function decline and changes to lung structure. It will investigate if this is mediated by inflammation, immune host response or elastin and collagen changes. It is an observational prospective cohort study aiming to recruit healthy controls, and people with asthma or COPD), and/or the menopause.

DETAILED DESCRIPTION:
The investigators are investigating the effect of oestrogen and oestrogen loss on the lungs. This is important to because lung diseases are a growing problem globally. In people suffering from Asthma and chronic obstructive pulmonary disease (COPD), women are more likely to die from lung disease than men. The researchers believe this global difference is due to sex hormones. Women have more oestrogen than men. Other studies have shown that oestrogen affects the lungs through the immune system. The researchers want to know the effect that oestrogen has on the lungs in people suffering from Asthma and COPD by comparing this to people with no lung disease. The researchers are also particularly interested in what happens at the point where women lose oestrogen naturally, which is the menopause. They want to understand the effect of oestrogen in younger women and compare this to women who have experienced the menopause. This is an observational study. Therefore, the participants will have a baseline visit and another subsequent visit (or multiple visits which are optional) and the researchers will compare the changes in their oestrogen levels, lung function and immune system response. To understand the differences mentioned above in the body we require samples and questionnaires to be filled out at face-to-face visits. All participants will be given the opportunity to opt into different streams of visits which vary between 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged > 18 years.
2. For female participants: pre-menopausal, peri-menopausal and post-menopausal women can all be included.
3. Participants willing and able to give informed consent for participation in the study.
4. Healthy controls <10 pack year history (participants without Asthma or COPD).

Exclusion Criteria:

1. Known or suspected current pulmonary tuberculosis, HIV (human immunodeficiency virus), Hepatitis B Virus, Hepatitis C Virus.
2. Alcohol or recreational drug abuse, is defined as when the use is harmful as per NHS definition.
3. History of psychiatric, medical, or surgical disorders.
4. Pregnant
5. Unable to provide written informed consent
6. History of advanced medical conditions with an expected prognosis of < 3 years.
7. Patients with a history of active cancer.
8. Patients on long term oxygen (ambulatory oxygen).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with physician-diagnosed disease (Asthma and/or COPD) or healthy controls
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Lung Function (FEV1 change from baseline) | Through study completion, minimum of 1 year
  Lung function measures the volume of air exhaled at specific time points during complete exhalation by force, which is preceded by a maximal inhalation.

SECONDARY OUTCOMES:
Oscillometry | Through study completion, minimum of 1 year
  Oscillometry is a technique that measures the mechanical impedance of the respiratory system, or how well the lungs are functioning.
The COPD Assessment Test (CAT) | Through study completion, minimum of 1 year
  The COPD Assessment Test (CAT) is a questionnaire for people with Chronic Obstructive Pulmonary Disease (COPD). It is designed to measure the impact of COPD on a person's life, and how this changes over time
Asthma Control Questionnaire (ACQ) | Through study completion, minimum of 1 year
  A simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment.
Asthma Quality of Life Questionnaire (AQLQ) | Through study completion, minimum of 1 year
  A disease-specific health-related quality of life instrument that taps both physical and emotional impact of disease. The instrument should not be confused with the measure developed by Marks GB and colleagues, which carries the same name.
EQ-5D-5L | Through study completion, minimum of 1 year
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
The Greene Climacteric Scale (GCS) | Through study completion, minimum of 1 year
  is a questionnaire that helps to determine the severity of menopausal symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, Principal Investigator — King's College London
Locations (1):
- Guys & St Thomas NHS Foundation Trust, London, United Kingdom